CLINICAL TRIAL: NCT06933758
Title: Temple Health Chest Initiative (THCI 2.0) - Lung Cancer Screening Project With COPD Detection
Brief Title: Temple Health Chest Initiative (THCI 2.0)
Status: Recruiting | Type: Observational
Sponsor: Temple University (Other)
Responsible Party: Sponsor
Other Study IDs: THCI 2.0 RESEARCH PLAN
Record Dates: First submitted 2025-01-22; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-01

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tomography, X-Ray Computed; Symptom Assessment

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pulmonary function testing: If the patient does have airflow obstruction (any severity) they will be contacted to complete additional questionnaires.
  Interventions: Diagnostic Test: Determine COPD prevalence utilizing spirometry along with CT scans and symptom assessments in the THCI lung cancer screening populatio

INTERVENTIONS:
Diagnostic Test: Determine COPD prevalence utilizing spirometry along with CT scans and symptom assessments in the THCI lung cancer screening populatio — Demonstrate utility of LDCT in COPD characterization Determine exacerbation risk and symptom burden in this patient population Determine the severity of COPD identified through this process Describe phenotypic characteristics including imaging analysis of THCI population Determine the suitability and acceptance of patients to participate in COPD clinical trials Determine the incidence of comorbid lung (ILA, bronchiectasis, pulmonary artery enlargement) and non-lung problems (cardiac and aortic calcifications, osteopenia/osteoporosis and for gut abnormalities) identified by LDCT in a patient population at risk for lung cancer and/or COPD Determine the correlation between clinical measurements and imaging biomarkers

SUMMARY:
Chronic obstructive pulmonary disease is highly prevalent globally, with considerable morbidity and mortality associated. In the US, it is the 4th leading cause of death, as well as contributing to significant costs on healthcare utilization including hospitalization. Population-based screening for COPD has not been recommended by the US Preventative Services Task Force (USPSTF). However, LDCT screening for lung cancer in patients aged 50- 80 with ≥ 20 pack year smoking has been shown to improve survival. COPD is highly prevalent within LCS programs, with estimated rates of obstructive lung function of up to 59% and evidence of emphysema on CT scan in around 70%.

DETAILED DESCRIPTION:
The rates of undiagnosed COPD are reported to be between 20 to 40% 1, 2, 3 with all GOLD stages of disease identified. Of those with no known diagnosis, up to 50% had symptoms consistent with COPD1. Currently, population-based screening is not recommended for COPD by the US Preventive Services Task Force (USPSTF)4. However, given the overlapping risk factors for COPD and lung cancer, there are existing opportunities to target identification of COPD within a high-risk group and build further understanding of the impact on outcomes of earlier diagnosis, phenotyping of disease and implementation of treatment. Screening for early lung cancer using low dose CT imaging also affords the opportunity to explore presence of comorbidities on images, such as presence and extent of emphysema and other lung parenchymal and airway abnormalities and coronary artery calcification. There is also an opportunity to explore the role of imaging biomarkers for COPD such as LAA and airway inflammation, in determining risk of disease progression through longitudinal observation.

ELIGIBILITY:
Inclusion Criteria:

* 50 to 80 years old
* Screened for early lung cancer using low dose CT imaging

Exclusion Criteria:

* Under 50; over 80 years old
* No lung cancer screening

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * 50 to 80 years old
  * screened for early lung cancer using low dose CT imaging
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
COPD Prevalence | 15 months
  Determine COPD prevalence utilizing < 0.7 FEV1/FVC plus evidence of emphysema by quantitated HRCT in the THCI lung cancer screening population.

SECONDARY OUTCOMES:
Severity of COPD | 15 months
  Determine the severity of COPD identified by FEV1 % predicted
Demographic Characteristics | 15 months
  Describe demographics characteristics of THCI population
Incidence of Comorbid Lung and Non-lung Problems | 15 months
  Determine the incidence of comorbid lung (ILA, bronchiectasis, pulmonary artery
  enlargement) and non-lung problems (cardiac and aortic calcifications,
  osteopenia/osteoporosis and for gut abnormalities) identified by LDCT in a patient
  population at risk for lung cancer and/or COPD

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Criner, MD, Principal Investigator — Temple University
Locations (1):
- Temple University Of the Commonwealth System of Higher Education, Philadelphia, Pennsylvania, United States